CLINICAL TRIAL: NCT02138682
Title: Validation of DaTscan for Detection of Parkinsonian Disease and Related Disorders Using Neuropathologically-confirmed Parkinson Disease From Human Brain Tissue
Brief Title: Validation of DaTscan for Detection of Parkinson Disease Related Disorders
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Wisconsin Institute for Neurologic and Sleep Disorders S.C. (Industry)
Collaborators: Wisconsin Parkinson Association (Unknown); Medical College of Wisconsin (Other); GE Healthcare (Industry)
Responsible Party: Principal Investigator, Paul Nausieda, Medical Director, Wisconsin Institute for Neurologic and Sleep Disorders S.C.
Other Study IDs: 12-DAT-014
Record Dates: First submitted 2014-04-24; First posted 2014-05-14 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Parkinson Disease; Movement Disorders
Keywords: DaT-SPECT scan; Parkinson's; Diagnostic
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Disease | interventions — ioflupane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fixed brain tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- l-123 Ioflupane: Study group includes those clinically diagnosed with Parkinson disease who are aged 75 and older who have agreed to donate brain tissue at time of death and are able to participate in the imaging scan process.
  Interventions: Drug: l-123 Ioflupane

INTERVENTIONS:
Drug: l-123 Ioflupane — 5 millicuries of Ioflupane
  Other Names: DaTscan

SUMMARY:
This investigator initiated trial is designed to measure the accuracy of diagnosis of Parkinson disease through the use of DaTscan. Currently, DaTscan is FDA approved to measure dopamine transporter densities in human tissue. This measurement can assist in distinguishing between Essential Tremor and Parkinsonian Syndromes (idiopathic Parkinson disease, Progressive Supranuclear Palsy, Multi Systems Atrophy, etc). This study will compare both clinical diagnosis of symptoms and the results of the scan to the pathological diagnosis received at time of death. Patients will be registered in the Parkinson Research Institute's brain donation program, receive a clinical diagnosis of Parkinson disease, have their brain scanned using DaTscan, and donate their tissue for research and autopsy purposes. The hypothesis of the study is that DaTscan will diagnosis Idiopathic Parkinson Disease as accurately as a clinician.

ELIGIBILITY:
Inclusion Criteria:

* aged 75 or older
* sporadic late onset Parkinson disease or one of its variants
* registered in tissue donation program

Exclusion Criteria:

* aged less than 75 years old
* mental status preventing neuroimaging or transportation to site
* inability to remain "relatively steady" during the scanning procedure

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Parkinson disease patients from Wisconsin Institute for Neurologic and Sleep Disorders, SC.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Consistency Between Diagnostic Procedures | Will be assessed upon receipt of autopsy report- time frame per patient is 24 months from enrollment.
  Consistency of diagnosis between: (1) clinical diagnosis, (2) scan results, and (3) pathological results.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Nausieda, MD, Principal Investigator — Wisconsin Institute for Neurologic and Sleep Disorders
Locations (2):
- United States (2):
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Wisconsin Institute for Neurologic and Sleep Disorders, SC, Milwaukee, Wisconsin